CLINICAL TRIAL: NCT04519138
Title: Safety and Efficacy of the Endodrill Model X Biopsy Instrument When Sampling Tumours in the Upper Gastrointestinal Tract
Brief Title: Investigation to Evaluate Safety and Efficacy of the Endodrill Model X Biopsy Instrument
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Bibb Instruments AB (Unknown); Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BIBB EDMX01
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Tumor Sampling
Keywords: Endoscope; Gastrointestinal; Image-Guided Biopsy; Fine-Needle; Medical device; Methods; Diagnosis
MeSH Terms: conditions — Disease | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Intervention Model Description: Both the Endodrill Model X device and the standard instrument are used on the same lesion and patient to evaluate both instruments and their functions under as similar circumstances as possible.
Masking Description: The order of the instruments to be used is blinded to the endoscopist until after the tumor has been visualized to avoid and minimize the influence of the choice of instrument of where the sample is taken. Closed envelopes prepared according to a randomization list stratified by site are available at each site. The envelope is opened by an assistant and not shown to the examiner until the tumor has been visualized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endodrill Model X (Experimental): Three consecutive samples will be taken using the Endodrill Model X instrument.
  Interventions: Device: Endodrill Model X
- Endoscopic ultrasound guided fine-needle aspiration/biopsy (Active Comparator): Three consecutive samples will be taken using the the standard method fine-needle aspiration/biopsy.
  Interventions: Device: Fine-needle aspiration/biopsy

INTERVENTIONS:
Device: Endodrill Model X — The investigational device Endodrill Model X is used for biopsy sampling in the upper gastrointestinal tract
  Arms: Endodrill Model X
Device: Fine-needle aspiration/biopsy — The standard method is used for biopsy sampling in the upper gastrointestinal tract
  Arms: Endoscopic ultrasound guided fine-needle aspiration/biopsy

SUMMARY:
This is an investigator led prospective open label investigation, performed at three clinics in Sweden, comparing the flexible endoscopic biopsy instrument Endodrill Model X with the standard sampling method endoscopic ultrasound fine needle aspiration/biopsy. Assessment of safety is the primary objective and performance is the secondary objective.

DETAILED DESCRIPTION:
The investigation will include 20 patients with lesions and suspected tumors in the stomach, esophagus or duodenum (upper small intestine). The investigation will consist of one visit with an endoscopic examination with sampling of an observed lesion or suspected tumor. Six biopsies will be collected from each patient, three consecutive samples using the Endodrill Model X instrument and three consecutive samples using the standard fine needle. The order of instruments to be used will be randomly assigned. The patient will be under observation for 2 hours after the procedure. Telephone follow-up will be performed 1 and 7 days after the examination. Visual confirmation of the biopsies size will be recorded at the examination. If the samples verify a tumor or not will be evaluated at Day 14 when the pathology report is concluded.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age at the day of inclusion
* Signed informed consent
* Submucosal tumor of the upper gastrointestinal tract with tumor size ≥ 10 mm, well localized by the endoscopic examination

Exclusion Criteria:

* Suspicion of vascular tumor (e.g. pulsating tumor)
* Ongoing treatment with anticoagulants (e.g. Warfarin)
* Ongoing treatment with immunosuppressive drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with pre-specified adverse events | 10 days
  Proportion of patients with one or more of the following: 1) non-intentional perforation of the sampled organ, 2) bleeding requiring open surgical intervention or treatment at an intensive care unit, 3) non-planned hospitalization for observation AND where the patient is not fully recovered within 10 days after the endoscopic examination

SECONDARY OUTCOMES:
Amount of visible biopsy material over or under 5 mm at endoscopy examination | Day 0 (day of biopsy)
  Visual confirmation of the biopsies size > 5 mm or not, will be recorded at the examination. Analysis will be performed at each hospitals department of pathology as all biopsy samples are routinely handled. A copy of the pathology report will recorded in the Contact Report Form (CRF) at day 14 when the study report for each patient is concluded

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Swahn, MD, PhD, Principal Investigator — Skane University hospital, Lund, Sweden
Locations (3):
- Sweden (3):
  - Linköping University Hospital, Linköping
  - Skane University Hospital, Lund
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No